CLINICAL TRIAL: NCT05184140
Title: MELISA Trial: Mapping sEntinel Lymph Node in Initial StAges of Ovarian Cancer
Brief Title: Mapping Sentinel Lymph Node in Initial Stages of Ovarian Cancer
Acronym: MELISA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Berta Diaz-Feijoo (Unknown); Aureli Torné (Unknown); Pilar Paredes (Unknown); Sergi Vidal-Sicart (Unknown); Ariel Glickman (Unknown); Pere Fusté (Unknown); Tiermes Marina (Unknown); Francisco Campos (Unknown)
Responsible Party: Principal Investigator, Núria Agustí, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCB/2021/0130
Record Dates: First submitted 2021-12-04; First posted 2022-01-11 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer; Sentinel Lymph Node
Keywords: Ovarian Cancer; Sentinel Lymph Node
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Controlled, prospective, descriptive
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adnexal mass with high suspicion of malignancy (Experimental): An ovarian lymphatic map will be performed in patients with adnexal masses suspected of malignancy. Sentinel node exeresis and a complete staging surgery (including pelvic and para-aortic lymphadenectomy) will be performed in patients with ovarian cancer confirmation including restaging surgeries.
  Interventions: Procedure: Sentinel node detection

INTERVENTIONS:
Procedure: Sentinel node detection — Injection of the radiotracer to infundibulo-pelvic and utero-ovarian ligament in patients with high suspicion of malignancy adnexal mass. Injection of green indocyanine r to infundibulo-pelvic and utero-ovarian stumps only in case of malignancy after the adnexectomy.
  Sentinel node exeresis and a complete staging surgery (including pelvic and para-aortic lymphadenectomy) will be performed in patients with ovarian cancer diagnosis.
  Other Names: Complete staging surgery

SUMMARY:
Epithelial ovarian cancer (EOC) diagnosed in the initial stage (stage I-II) require complete staging surgery to histologically assess the possible existence of peritoneal or lymph node disease.

Systematic pelvic and paraaortic lymphadenectomy in stage I-II EOC is essential since confirming the presence of lymph node metastases means re-staging the disease as stage III. This change of stage has important prognostic and therapeutic implications. However, the lymph node involvement rate is around 10-30% (average of 15%). Systematic pelvic and para-aortic lymphadenectomy carries a risk of intraoperative complications, as well as longer operative time, postoperative complications and longer hospital stay. Moreover, by now there is no evidence suggesting a possible therapeutic value.

The sentinel lymph node (SLN) detects the first level of lymph node drainage. The absence of metastases in the SLN predicts the absence of tumor infiltration of the rest of lymph nodes of the same anatomical region and allows to safely avoid lymphadenectomy and its associated morbidity. In addition, the exhaustive evaluation of the SLN by ultrastaging and immunohistochemical study allows to increase the detection of microscopic disease.

Sentinel lymph node (SLN) biopsy, implemented in clinical practice in other gynecological tumors (breast, vulva, cervix or endometrium), has been studied very little in the initial ovarian epithelial cancer. Unlike other gynecological tumors, there are multiple anatomical and technical aspects that largely explain this lack of information. The double ovarian vascularization that accompanies lymphatic drainage explains this higher complexity. Therefore, at the present time, the detection of SLN in the initial EOC remains an experimental area without applicability in clinical practice. There are multiple doubts and issues to be resolved regarding the different tracers, the site and time injection and the actual accuracy of the SLN versus the lymphadenectomy.

DETAILED DESCRIPTION:
The objective of this study is to know the lymphatic drainage and, if the lesion is malignant, remove the sentinel lymph nodes to know if it can predict the involvement of the remaining lymph nodes to assess the possible applicability of SLN in clinical practice.

Study design:

1. Evaluation of the ovarian lymphatic map: injection of radiotracer (99mTc-nanocolloid albumin) in patients with a diagnosis of adnexal mass with high suspicion of malignancy. Intraoperative lymphogammagraphy will be performed using a portable gammacamera. Patients with a delayed diagnosis of ovarian cancer who are candidates to undergo a re-staging surgery will be included.
2. After the adnexectomy a frozen section will be performed to confirm the diagnosis of malignancy and then the ICG (Indocyanine green) tracer will be injected. Since the spread and persistence of the ICG in the lymph nodes is rapid, this tracer will be injected only after confirmation of EOC. Simultaneous screening with a gammadetector probe and NIR (near-infrared spectrum) camera will be used to proceed to the detection of SLN according to the lymphatic map previously.
3. Ultrastaging of the SLN by applying hematoxylin and eosin staining (H&E) and, in the absence of metastatic disease, evaluation by immunohistochemistry with cytokeratin AE1: AE3.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of adnexal mass with high suspicion of malignancy and frozen section examination will undergo the lymphatic map with a radiotracer.
* Patients with intraoperative diagnosis of epithelial ovarian cancer will undergo the SLN exeresis with two tracers.
* Patients with a delayed diagnosis of epithelial ovarian cancer who are candidates to undergo a re-staging surgery will undergo the SLN exeresis with two tracers.

Exclusion Criteria:

* Advanced ovarian cancer (FIGO III/IV)
* Patients <18 years
* Pregnancy or lactation
* Previous vascular surgery (cava, aorta, iliac vessels), lymphadenectomy (pelvic or paraortic) or radiotherapy (pelvic or paraortic field)
* Severe adherent syndrome that prevents tracer injection
* The SLN technique will not be performed in case of benign ovarian tumor in the frozen section or borderline tumor (since in these cases there is no clinical indication of performing a lymphadenectomy)
* Non-operable patient
* Previous adverse events to the radiotracer or ICG

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Detection rate of sentinel node technique | Through study completion, an average of 2 years
  Detection of SLN in initial epithelial ovarian cancer by assessing the concordance of the result between the lymph node metastases and the lymphadenectomy

SECONDARY OUTCOMES:
Tracer specific detection rate | 2 years
  To know the global and specific SLN identification rate, depending on the type of tracer used.
Tracer-related adverse events | 1 month
  The number of patients with tracer-related adverse events
False negative rate and negative predictive value | 2 years
  Evaluate the existence of false negatives in metastatic involvement of the SLN and negative predictive value
Anatomical location of the sentinel lymph node | 2 years
  The aortic and pelvic region will be divided 13 regions
Detection rate of gamma-camera, gamma-probe and Infrared fluorescence camera | 2 years
  Evaluate the performance of intraoperative lymphoscintigraphy with gamma-camera, gamma-probe and Infrared fluorescence camera in the visualization of the ovarian lymphatic map.
Surgical time extension performing SLN technique | 2 years
  Evaluate the time it takes to perform the SLN technique
Anatomopathological ultrastaging examination of the sentinel lymph node | 2 years
  Evaluate if ultrastaging of the SLN improves the detection of micrometastases compared to conventional histology. Ultrastaging protocol will be performed, consisting of two consecutive histological sections (4 μm thick) obtained at regular intervals of 150 μm, performing 4 levels of each paraffin block. The first section will be stained with H&E and the second section will be stained immunohistochemically with an AE1-AE3 anti-keratin antibody (Dako®).

OTHER OUTCOMES:
Evaluation of sentinel lymph node technique | Through study completion, an average of 2 years
  To check the ovarian lymphatic drainage in patients with suspected malignant adnexal masses

CONTACTS AND LOCATIONS:
Overall Officials: Aureli Torné, PhD, Study Director — Hospital Clinic of Barcelona; Berta Díaz-Feijóo, PhD, Study Director — Hospital Clinic of Barcelona
Locations (1):
- Núria Agustí Garcia, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared only with those making official request to the study investigator
Supporting Information: Study Protocol, ICF
Time Frame: The data will become available One year after publication, and they will be available for 6 months.
Access Criteria: Direct request to the study PI

REFERENCES:
- See also: Sentinel lymph node mapping in early-stage ovarian cancer: surgical technique in 10 steps — http://dx.doi.org/10.1136/ijgc-2022-003420